CLINICAL TRIAL: NCT00156000
Title: Fetal Fibronectin (fFN) and Salivary Estriol (E3) in the Prediction of Preterm Birth in Women With Twin Pregnancies Receiving 17-Alpha-Hydroxyprogesterone Caproate or Placebo
Brief Title: fFN & E3 in the Prediction of PTB in Women With Twin Pregnancies Receiving 17OHP or Placebo
Status: Withdrawn | Type: Observational
Why Stopped: This study was stopped because of insufficient enrollment.
Sponsor: Obstetrix Medical Group (Industry)
Collaborators: Adeza Biomedical (Industry)
Responsible Party: Sponsor
Organization: Pediatrix (Other)
Other Study IDs: OBX0048.2
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Preterm Delivery; Preterm Birth
Keywords: Preterm Delivery; Multifetal pregnancy; Preterm Birth; 17-alpha Hydroxyprogesterone Caproate; Markers of Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Fetal Fibronectin — fFN test done during pregnancy
  Other Names: fFN
Device: Salivary Estriol — Salivary Estriol done during pregnancy
  Other Names: SalEst

SUMMARY:
Among women with a twin pregnancy, currently enrolled in a study in which they are receiving weekly injections of 17-alpha-hydroxyprogesterone caproate verses placebo injections, fetal fibronectin (fFN) and salivary estriol (E3 ) will identify the following.

1. Women at increased risk for preterm delivery.
2. A subpopulation, among those receiving the active drug, who may respond to progesterone.

If fFN and/or E3 identify a population of patients who respond to progesterone, these diagnostic tests may define women who may or may not be good candidates for progesterone therapy.

DETAILED DESCRIPTION:
Preterm birth occurs in approximately 12% of all pregnancies in the United States and is the leading cause of neonatal morbidity and mortality. Despite extensive efforts the preterm birth rate has risen 25% in the United States over the last two decades. Women with multi-fetal pregnancies are at especially high risk of preterm birth. About half of twin pregnancies and almost all triplet pregnancies result in preterm birth. Thus, women with multi-fetal gestations appear to be a group that would benefit most from a screening intervention to determine those pregnancies at greatest risk for preterm birth. Currently, two biochemical, diagnostic tests for preterm birth are approved by the FDA: fetal fibronectin and salivary estriol testing. Recent studies have shown that weekly administration of 17-alpha-hydroxyprogesterone significantly reduced preterm delivery in singleton pregnancies. The proposed study will assist in the assessment of women who will benefit most from progesterone injections by clarifying it's mechanism of action through the evaluation of serial fFN and E3 samples in a subset of women currently enrolled in a multi-center trial evaluating 17-alpha-hydroxyprogesterone caproate in twin and triplet pregnancies.

This is a prospective observational study following the results of serial fetal fibronectin and salivary estriol samples in a subpopulation of women with twin pregnancies currently enrolled in a primary trial of weekly injections of 17-alpha-hydroxyprogesterone caproate versus placebo injections. Subjects will be recruited from a large perinatology practice consisting of four outpatient clinics in the Phoenix metropolitan area.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with twin pregnancies currently participating in the ongoing IRB approved multicenter trial entitled 17-Alpha-Hydroxyprogesterone Caproate for Reduction of Neonatal Morbidity due to Preterm Birth in Twin and Triplet Pregnancy.
2. GA at time of enrollment between 16w0d weeks gestation and 23w6d gestation)
3. Maternal age 18 years or older
4. Intact amniotic membranes
5. Investigator believes patient will be reliable with follow-up visits and believes that delivery data & neonatal data are likely to be available.
6. Subject has voluntarily signed and dated an IRB approved informed consent form prior to any participation in the study

Exclusion Criteria:

1. Symptomatic uterine contractions at time of enrollment
2. Placenta previa
3. Abruptio placenta
4. Severe preeclampsia
5. Digital examination within 24 hours prior to the fFN sample collection
6. Vaginal intercourse within 24 hours prior to the fFN sample collection
7. Transvaginal ultrasound or vaginal speculum exam within 24 hours prior to fFN sample collection
8. Amniocentesis within 24 hours prior to fFN sample collection
9. Moderate or gross vaginal bleeding at the time of fFN sample collection
10. Cervical cerclage
11. Advanced cervical dilatation ≥ 3 cm

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women (Twins or Triplets) already enrolled in the Obstetrix Clinical Trial " Progesterone for prevention of PTB in twin and triplet pregnancies"
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2005-08; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Maurel, RN, MSN, CNS, Study Director — Obstetrix Medical Group, Inc.; Richard Lee, Principal Investigator — Obstetrix Medical Group, Inc.
Locations (2):
- United States (2):
  - Desert Good Samaritan Hospital, Mesa, Arizona
  - Banner Good Sammaritan Hospital, Phoenix, Arizona

REFERENCES:
- [Background] Goldenberg RL, Mercer BM, Meis PJ, Copper RL, Das A, McNellis D. The preterm prediction study: fetal fibronectin testing and spontaneous preterm birth. NICHD Maternal Fetal Medicine Units Network. Obstet Gynecol. 1996 May;87(5 Pt 1):643-8. doi: 10.1016/0029-7844(96)00035-x. PMID 8677060
- [Background] Darne J, McGarrigle HH, Lachelin GC. Increased saliva oestriol to progesterone ratio before preterm delivery: a possible predictor for preterm labor? Br Med J (Clin Res Ed). 1987 Jan 31;294(6567):270-2. doi: 10.1136/bmj.294.6567.270. PMID 3101838